CLINICAL TRIAL: NCT03348371
Title: The Effects of Orally Ethanol vs. Isoethanolaemic i.v. Infusion of Ethanol on Intestinal Permeability and Gut Hormones
Brief Title: The Effects of Ethanol on Intestinal Permeability and Gut Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Amalie Lanng, BA, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AlcoGut
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Insulin Resistance; Ethanol; Incretin Effect
Keywords: Incretin effect; Ethanol
MeSH Terms: conditions — Insulin Resistance | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral day (Experimental): Participant receive ethanol orally
  Interventions: Other: Ethanol
- i.v. infusion day (Experimental): Participant receive ethanol in an i.v. infusion
  Interventions: Other: Ethanol

INTERVENTIONS:
Other: Ethanol — The intervention is two different administrationforms of ethanol, orally and i.v.

SUMMARY:
The aime of this study is to envsitigate if ethanol has an incretin effect. This is done by administration of ethanol orally vs. an isoethanolaemic i.v. infusion of ethanol.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male between 20 and 50 years of age
* Body mass index (BMI) between 19 and 25 kg/m2
* Weekly alcohol intake of less than 14 units of alcohol (of 12 g)
* Normal fasting plasma glucose concentration (i.e. <6 mmol/l) and normal glycated haemoglobin A1c (HbA1c) (i.e. ≤42 mmol/mol)
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* First-degree relatives with diabetes and/or liver disease
* Liver disease or other alcohol-related diseases, diabetes mellitus
* Liver disease (serum ALAT and/or serum ASAT >2 × normal values)
* Nephropathy (serum creatinine above normal range and/or albuminuria)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Serum insulin level | 2 month
  difference in serum insulin level between the two administration forms

IPD SHARING:
Plan to Share IPD: No